CLINICAL TRIAL: NCT06853496
Title: Investigator-initiated Phase I Study of a Tankyrase Inhibitor RK-582 for Patients With Unresectable Metastatic Colorectal Cancer
Brief Title: Study of a Tankyrase Inhibitor RK-582 for Patients With Unresectable Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eiji Shinozaki (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Sponsor-Investigator, Eiji Shinozaki, Vice Director of Gastroenterological Chemotherapy Department, Japanese Foundation for Cancer Research
Organization: Japanese Foundation for Cancer Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RK582CRCPI; jRCT2031240702 (Registry Identifier: Japan Registy of Clinical Trials)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-02

CONDITIONS: Unresectable Colorectal Neoplasm Metastasis
Keywords: colorectal neoplasm; colorectal cancer; tankyrase inhibitor
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RK-582 (Experimental)
  Interventions: Drug: RK-582

INTERVENTIONS:
Drug: RK-582 — Dosing Frequency:
  Do single dose of RK-582 at the dose level specified for the cohort. Seven days after the first dose, Start repeated daily dose and continue until discontinuation criteria were met.
  Dose level per dose:
  Dose Level 1: 5 mg BID Dose level 2: 10 mg QD Dose level 3: 20 mg QD Dose level 4: 40 mg QD Dose Level 5: 60 mg QD Dose Level 6: 80 mg QD Dose Level 7: 100 mg QD Dose Level 8: 200 mg QD

SUMMARY:
Tankyrase, the fifth and sixth members of the poly(ADP-ribose) polymerase (PARP) family (PARP-5a/b), is responsible for poly(ADP-ribosyl)ation (PARylation), and was originally identified as a factor that promotes the function of telomerase, an enzyme that elongates telomeres. Subsequently, it was reported that tankyrase enhances Wnt/beta-catenin signaling by PARylation and subsequent degradation of AXIN, a negative regulator of Wnt/beta-catenin signaling, suggesting that tankyrase inhibitors may be a new treatment for colorectal cancer.

RK-582 was discovered through lead optimization from a tankyrase inhibitor that suppresses the growth of human colorectal cancer cells. It was confirmed that RK-582 selectively inhibited tankyrase among the PARP family enzymes, suppressed the growth of Wnt/beta-catenin signal-dependent human colorectal cancer cells at both the levels of cultured cells and xenograft tumors in immunodeficient mice, and accumulated AXIN to decrease beta-catenin and downregulate the target gene expression as pharmacodynamic biomarkers.

Based on these findings, RK-582 is thought to have potential as a new treatment for colorectal cancer patients. At present, however, the efficacy and safety of RK-582 in humans have not been confirmed. Thus, this clinical trial is conducted with the aim of investigating the tolerability and safety of RK-582 for patients with unresectable advanced or recurrent colorectal cancer as a first-in-human trial, in which RK-582 is administered to humans for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically diagnosed colorectal cancer
* Patients who are refractory or intolerant to standard treatment for unresectable advanced or recurrent colorectal cancer
* Patients with measurable disease according to RECIST guideline ver 1.1
* Patients who are able to take capsules orally

Exclusion Criteria:

* Patients with clinically relevant gastrointestinal, hepatic, musculoskeletal, respiratory, cerebral/cardiovascular, hematologic, oncologic, endocrine, immunologic, psychiatric, neurologic, or genitourinary diseases, or patients with conditions that are judged to threaten the safety of the participant or to affect the outcome of this clinical trial by the investigators
* Patients with medical history of interstitial lung disease
* Patients with chronic nausea, vomiting or diarrhea that may interfere with oral administration of the investigational drug
* Patients with pulmonary embolism or central deep vein thrombosis.
* Patients receiving treatment with strong CYP3A4 inhibitors or inducers.
* Patients diagnosed and treated for osteoporosis or patients with a bone mineral density of less than T-score -2.5 at the time of screening
* Patients with obvious bone metastases in the long bones, vertebrae, or other parts of the leg where gravity is applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of dose-limiting toxicity | 35 days after the first dose of RK-582
Number of participants with adverse events as assessed by CTCAE v5.0 | Approximately 1 year after the first dose of RK-582

SECONDARY OUTCOMES:
Area under the curve (AUC) after single or repeated dosing | 22 days after the first dose of RK-582
Maximum plasma concentration (Cmax) after single or repeated dosing | 22 days after the first dose of RK-582
Maximum concentration time (Tmax) after single or repeated dosing | 22 days after the first dose of RK-582
Elimination rate constant (kel) after single or repeated dosing | 22 days after the first dose of RK-582
Elimination half-life (t1/2) after single or repeated dosing | 22 days after the first dose of RK-582
Apparent total body clearance (CLtot/F) after single or repeated dosing | 22 days after the first dose of RK-582
Apparent volume of distribution (Vd/F) after single or repeated dosing | 22 days after the first dose of RK-582
Objective response rate based on investigator's judgment as assessed by RECIST guideline ver. 1.1 | Approximately 1 year after the first dose of RK-582
Percentage of subjects who achieved a complete or partial response on the best overall response as assessed by RECIST guideline ver. 1.1 | Approximately 1 year after the first dose of RK-582
Duration of response as assessed by RECIST guideline ver. 1.1 | Approximately 1 year after the first dose of RK-582
Disease control rate as assessed by RECIST guideline ver. 1.1 | Approximately 1 year after the first dose of RK-582
Time to response as assessed by RECIST guideline ver. 1.1 | Approximately 1 year after the first dose of RK-582
Progression-free survival as assessed by RECIST guideline ver. 1.1 | Approximately 1 year after the first dose of RK-582
Overall survival | Approximately 30 months after the first dose of RK-582

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Yamaguchi, Study Chair — Cancer Institute Hospital of JFCR
Locations (1):
- Cancer Institute Hospital of JFCR, Koto-ku, Tokyo, Japan